CLINICAL TRIAL: NCT00621335
Title: A 12- Week Investigator Masked, Parallel Comparison of Tolerability of Combigan and Cosopt in the Treatment of Open Angle Glaucoma or Ocular Hypertension
Brief Title: A Investigator Masked Parallel Comparison of Tolerability of Combigan and Cosopt
Acronym: CICOM1010
Status: Completed | Type: Observational
Sponsor: DBYAN Medicine Professional Corporation (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Dr. David Yan, Dr. David Yan M.D, F.R.C.S (c), DBYAN Medicine Professional Corporation
Other Study IDs: CICOM 1010
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Open angle glaucoma; Ocular hypertension; Parallel comparison; Combigan; Cosopt
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this research study is to compare the tolerability and effectiveness of Combigan(brimonidine tartrate/timolol maleate) and Cosopt (dorzolamide hydrochloride)in the treatment of open angle glaucoma or ocular hypertension.

DETAILED DESCRIPTION:
Patients between the ages of 40 to 90 years of age, that have been diagnosed with open angle glaucoma or ocular hypertension,including pseudo-exfoliation and pigmentary glaucoma with definitive glaucomatous optic disk cupping and/or glaucomatous visual field loss, who have been receiving a stable treatment regime for at least 4 weeks prior to the study initiation, with a Cosopt mono or a Prostaglandin + Cosopt combination are to be included in the study.Patients must have an IOP between 16 and 32 mmHg, with no readings above 35 mmHg at baseline.

Patients with any other form of glaucoma other than primary open angle glaucoma, with a gonioscopy measured angle grade of less than 2, with a visual field defect not of glaucomatous origen and previous cyclodestructive procedures will be excluded.The use of ocular non steroidal and anti-inflammatory topical agents which inhibit cyclooxygenase and prostaglandin analog synthesis,the use of glucocorticoid therapy, and hypersensitivity to any of the study components also precludes involvement in the study. Any ocular laser therapy within the past three months, ocular inflammation or infection in the past three months or any history of trauma in the last six months will also exclude enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* open angle glaucoma or ocular hypertension including pseudo-exfoliation and pigmentary glaucoma
* definitive glaucomatous optic disk cupping and/or glaucomatous visual field loss
* a stable treatment regime for at least 4 weeks prior to the study initiation, with a Cosopt mono or a Prostaglandin + Cosopt combination
* an IOP between 16 and 32 mmHg, with no readings above 35 mmHg at baseline

Exclusion Criteria:

* any other form of glaucoma other than primary open angle glaucoma
* a gonioscopy measured angle grade of less than 2
* a visual field defect not of glaucomatous origen
* previous history of cyclodestructive procedures
* the use of ocular non steroidal and anti-inflammatory topical agent that inhibit cyclooxygenase and prostaglandin analog synthesis
* the use of glucocorticoid therapy
* hypersensitivity to any of the study components
* any ocular laser therapy within the past three months
* ocular inflammation or infection in the past three months
* any history of trauma in the last six months

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2007-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Comparison of the tolerability and effectiveness of Combigan and Cosopt in the treatment of open angle glaucoma or ocular hypertension | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Yan, M.D., Principal Investigator — University of Toronto
Locations (1):
- Ophthalmic Consultants Centres, Mississauga, Ontario, Canada